CLINICAL TRIAL: NCT01248377
Title: The Results of Skin Testing and The Detection of Cytokine Secretion From Drug Specific Peripheral Blood Mononuclear Cells Using ELISPOT Assay in the Diagnosis of Nonimmediate Reactions to Cephalosporins
Brief Title: Skin Testing and ELISPOT Assay in Patients With a History of Non-Immediate Reactions to Cephalosporins
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jettanong Klaewsongkram, Faculty of Medicine, Department of Medicine, Chulalongkorn University
Other Study IDs: Chula-ARC 002/10
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cephalosporin Allergy; Non-immediate Drug Reactions
Keywords: Cephalosporins; Drug hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Skin Tests; Patch Tests; Intradermal Tests; Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMCs and serum will be collected for further analysis, if indicated
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cephalosporins allergic patients
  Interventions: Procedure: Skin tests and ELISPOT assay

INTERVENTIONS:
Procedure: Skin tests and ELISPOT assay — Patch test and/or intradermal test will be performed in patients as well as cytokine secretions from PBMCs will be analyzed by ELISPOT assay
  Other Names: Patch test; Intradermal test; ELISPOT

SUMMARY:
This study aims to compare the results of skin testing and ELISPOT assay in patients with a history of non-immediate reactions to cephalosporins

DETAILED DESCRIPTION:
Patients with a history of non-immediate reactions to cephalosporins will be tested by patch test and/or intradermal test. Peripheral blood mononuclear cells will be collected to analyzed cytokine secretions by ELISPOT assay

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of non-immediate hypersensitivity reactions to cephalosporins
2. At least 18 years of age

Exclusion Criteria:

1. Suffering from severe systemic disease/ in bad health
2. Being pregnant
3. Patients with a history of immediate reactions to cephalosporin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of non-immediate hypersensitivity reactions to cephalosporins
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The skin testing results of Cephalosporin skin test compared to ELISPOT assay | 1 year

SECONDARY OUTCOMES:
The result of cross reactivity between Cephalosporins and other Betalactams determined by skin testing and ELISPOT assay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Tanvarasethee B, Buranapraditkun S, Klaewsongkram J. The potential of using enzyme-linked immunospot to diagnose cephalosporin-induced maculopapular exanthems. Acta Derm Venereol. 2013 Jan;93(1):66-9. doi: 10.2340/00015555-1386. PMID 22722755